CLINICAL TRIAL: NCT04541602
Title: Value of Neuromuscular Ultrasound and Blood Biomarkers for the Detection, Monitoring and Prognostication of Neuromuscular Complications in Critically Ill Patients: a Prospective Single-center Observational Study
Brief Title: Detection of Neuromuscular Complications in Critically Ill Patients
Acronym: NMCiCIP
Status: Terminated | Type: Observational
Why Stopped: PI and the majority of the study team left institution.
Sponsor: University of Rostock (Other)
Responsible Party: Principal Investigator, Dr. Johannes Ehler, MD, PD Dr. med. Johannes Ehler, MD, University of Rostock
Other Study IDs: NMCiCIP
Record Dates: First submitted 2020-09-01; First posted 2020-09-09 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Critical Illness; Dysphagia; Intensive Care Unit Acquired Weakness; Neuromuscular Diseases
MeSH Terms: conditions — Critical Illness; Deglutition Disorders; Neuromuscular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Dysphagia-positive: * critically ill patients more than 17 years of age
  * matching study inclusion criteria
  * confirmed newly acquired swallowing dysfunction using FEES at study day 10 or later
  * ICU-AW positive (MRC-ss <48) or ICU-AW negative (MRC-ss ≥48)
- Dysphagia-negative: * critically ill patients more than 17 years of age
  * matching study inclusion criteria
  * newly acquired swallowing dysfunction ruled out using FEES at study day 10 or later
  * ICU-AW positive (MRC-ss <48) or ICU-AW negative (MRC-ss ≥48)
- Controls: * healthy volunteers without any neuromuscular disease
  * swallowing dysfunction ruled out using FEES

SUMMARY:
Dysphagia and the intensive care unit-acquired weakness (ICU-AW) are common and outcome-relevant neuromuscular complications in critically ill patients, especially after prolonged mechanical ventilation, sepsis and multi-organ failure. However, the impact of these two complications on the clinical course of critically ill patients needs further investigation.

Furthermore, the standard diagnostic procedure to detect and grade the acquired dysphagia using the fiberoptic endoscopic evaluation of swallowing (FEES) and the Medical Research Council sum score (MRC-ss) to detect ICU-AW are time-consuming and strongly dependent on patient compliance. An early and easy-to-use detection of these neuromuscular complications is currently difficult to be achieved in this patient population.

Neuromuscular ultrasound (NMUS) and the measurement of neuromuscular damage blood biomarkers became increasingly interesting for clinical researchers in the recent years due to their broad availability and their simple and non-invasive application. However, the value of these new diagnostic tests to evaluate dysphagia and ICU-AW needs to be verified.

DETAILED DESCRIPTION:
In this single-center observational study the investigators aim to evaluate neuromuscular ultrasound and blood biomarkers of neuromuscular damage as innovative diagnostic features for the detection, monitoring and prognostication of dysphagia and ICU-AW in critically ill patients. A detailed neurological examination, NMUS as well as blood biomarker measurements (e.g. Myl3, TNNI1, FABP-3) will be longitudinally performed at study day 1 (day of study inclusion), day 3, day 10 and day 17 after study inclusion. The neurological examination comprises the use of validated scales (GCS, RASS, mRS) and scores (MRC-ss) to assess consciousness, neurological disability and muscle strength as well as the the examination of the reflex status. Using a standardized in-house NMUS protocol the facial (masseter muscle), submental (digastricus muscle, mylohyoid muscle), cervical (sternocleidomastoid muscle) and extremity muscles (biceps brachii, brachiradialis, quadriceps femoris, tibialis anterior) as well as the vagus nerve will be assessed repeatedly. Additionally, a FEES as the current gold standard diagnostic for dysphagia will be performed at study day 10 or as soon as possible (depending on the ability of the patient to cooperate with the examiner) after study day 10 to detect and grade the dysphagia.

All study participants will be reevaluated at day 90 after study inclusion with regard to functional disability and survival.

Furthermore, healthy volunteers will be recruited and assessed in the same way as patients including a clinical examination, NMUS, laboratory testing and FEES.

The investigators hypothezise that:

* acquired dysphagia due to critical illness (not caused by central nervous system damage) is more likely in patients with ICU-AW
* the outcome in patients with a combination of ICU-AW and dysphagia is worse compared to patients with only one of these entities
* NMUS is able to detect and monitor dysphagia and ICU-AW in critically ill patients who are at risk of neuromuscular dysfunction
* specific blood biomarker levels correlate with the severity of neuromuscular impairment and are of value to identify patients with ICU-AW and acquired dysphagia

ELIGIBILITY:
Inclusion Criteria:

* adult patients above 17 years of age
* Sequential organ failure assessment (SOFA) score ≥8 within the first two days after ICU admission
* invasive mechanical ventilation ≥48 hours

Exclusion Criteria:

* no written informed consent from patient or legal representative
* participation in another interventional study
* patient transfer from another hospital (>1 day hospital stay)
* preexisting swallowing disorder or disease of the larynx, pharynx or esophagus
* previous surgery of the larynx, pharynx, esophagus or maxillofacial surgery
* preexisting neuromuscular diseases
* preexisting central nervous system diseases (stroke, hemorrhage, tumor, traumatic brain injury, brain surgery, epilepsy, hydrocephalus)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the intensive care units of the study center will be screened for study eligibility according to the inclusion and exclusion criteria. Additionally, healthy volunteers will be recruited to participate as controls.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2024-12-08 (Actual); Study Completion 2024-12-08 (Actual)

PRIMARY OUTCOMES:
Incidence of sensomotory dysphagia in critically ill patients with and without intensive care unit-acquired weakness as well as controls | Day 90
  Assessment of dysphagia and ICU-AW using validated diagnostics (FEES, NMUS) and scores (MRC-ss)
Changes in ultrasonographic parameters between patients with and without newly acquired sensomotory dysphagia as well as controls | Change from baseline ultrasound parameters at day 17
  NMUS protocol performed at study days 1, 3, 10 and 17
Change in neuromuscular damage blood biomarker levels in critically ill patients with and without newly acquired sensomotory dysphagia as well as controls | Change from baseline parameters at day 17
  Specific blood biomarker levels (e.g. TNNI1, FABP-3) measured at study days 1, 3, 10 and 17

SECONDARY OUTCOMES:
Quality of life in patients with and without neuromuscular complications after hospital discharge | Day 90
  Assessment of the overall quality of life using validated tests [e.g. Modified Rankin Scale with a range from 0 (no symptoms) to 6 (dead)]
Length of hospital stay comparing critically ill patients with and without neuromuscular complications | 1 year
  Cumulative days in hospital
Survival in critically ill patients with and without neuromuscular complications | Day 28
  Survival after 28 days
Survival in critically ill patients with and without neuromuscular complications | Day 90
  Survival after 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Felix Klawitter, MD, Principal Investigator — University of Rostock; Johannes Ehler, MD, Principal Investigator — University of Rostock
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine, University Medical Center Rostock, Rostock, Mecklenburg-Vorpommern, Germany

IPD SHARING:
Plan to Share IPD: No